CLINICAL TRIAL: NCT01038921
Title: Melatonin Supplementation and the Metabolic Syndrome: A Phase II Crossover Design Clinical Trial
Brief Title: Melatonin and the Metabolic Syndrome
Acronym: MetSyn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael Kutner, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00014784; R21AT004220-01A2 (NIH)
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Metabolic Syndrome
Keywords: Blood Pressure; Glucose levels; HDL levels; Triglyceride levels; Waist Circumference
MeSH Terms: conditions — Metabolic Syndrome | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental): Melatonin 8mg one hour before bedtime for 10 weeks
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo administered 1 hour before bedtime for 10 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 8 mg dose of Melatonin
  Arms: Melatonin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This trial seeks to compare the effects of melatonin supplementation versus placebo in subjects with the metabolic syndrome.

DETAILED DESCRIPTION:
The primary purpose of this Phase II crossover design trial is to examine the safety and efficacy of 8mg of melatonin taken one hour before bedtime compared to a placebo treatment to improve at least one of the five components associated with the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-79 years.
2. Diagnosed with metabolic syndrome according to AdenosineTriphosphate-III criteria.
3. Availability for six months after enrolling in the study.

Exclusion Criteria:

1. Inability to understand informed consent and to cooperate with study procedures.
2. Supplemental intake of melatonin.
3. Current smoking.
4. Current use of calcium channel blockers.
5. Current, planned, or recent (12 months) participation in another clinical trial.
6. Women who are pregnant, breast-feeding, attempting conception, or planning to attempt conception over the next 6 months.
7. Presence of any of the following diagnosed health conditions:

   * Active malignancy other than nonmelanoma skin cancer (current therapy for this malignancy,diagnosis within five years of enrollment, recurrence within five years of enrollment, or metastasis)
   * Uncontrolled hypothyroidism or hyperthyroidism
   * Recent (< 1 year ago) history of heart attack, bypass surgery, angioplasty, or stroke
   * Heart failure (New York Heart Association functional class 3 or 4)
   * On renal dialysis
   * Immunosuppressive therapy (systemic corticosteroids, azathioprine, methotrexate, cyclophosphamide,
   * etc.) or an immunodeficiency syndrome
   * Narcotic or alcohol dependence
   * Obstructive sleep apnea (OSA) , defined either by previous diagnosis (with or without use of nasal CPAP), or by a score of 0.80 or higher on the MAP (Multivariate Apnea Prediction), a validated screening algorithm with high positive and negative predictive value for identifying OSA.
8. Shift-workers.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Kutner, PhD, Principal Investigator — Emory University; Abinav Goyal, M.D., Study Director — Emory University
Locations (2):
- United States (2):
  - Emory Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

REFERENCES:
- [Derived] Goyal A, Terry PD, Superak HM, Nell-Dybdahl CL, Chowdhury R, Phillips LS, Kutner MH. Melatonin supplementation to treat the metabolic syndrome: a randomized controlled trial. Diabetol Metab Syndr. 2014 Nov 18;6:124. doi: 10.1186/1758-5996-6-124. eCollection 2014. PMID 25937837
- See also: Published manuscript describing the study design of Melatonin Supplementation and the Metabolic Syndrone — http://www.dovepress.com/design-and-rationale-of-a-randomized-controlled-trial-of-melatonin-sup-peer-reviewed-article-OAJCT-recommendation1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from 05/24/2010 through 12/15/2011. Recruitment was from subjects from the "Screening for Impaired Glucose Tolerance: Glucose Challenge versus Predictive Model NIH study R18DK066204,from Preventive Cardiology Clinic at Emory University Clinic and from advertisements placed on the campus of the Emory Clinic
Pre-assignment Details: One week run in period on placebo. Six week washout period between crossover.
Groups:
- Melatonin: Cross-over design with subject receiving either Melatonin First and Placebo Second or Placebo First and Melatonin Second
- Placebo: Cross-over design with subjects receiving either Placebo First and Melatonin Second or Melatonin First and Placebo Second
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 19 (19 subjects received melatonin first(10 weeks), washout (6 weeks), placebo second (10 weeks)) | 20 (20 subjects received placebo first (10 weeks), washout (6 weeks), melatonin second ( 10 weeks))
Completed | 17 (2 subjects withdrew) | 20
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Expected to enroll 40 subjects but only randomized 39 subjects
Groups:
- Melatonin First: Cross-over design with subjects receiving Melatonin First
- Placebo First: Cross-over design with subjects receiving Placebo First
- Total: Total of all reporting groups
Arm/Group | Melatonin First | Placebo First | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 18 | 33
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.6) | 57.6 (10.1) | 58.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 10 | 12 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants] — Melatonin First Placebo First Caucasian 13 11 African American 6 7 Other 0 2
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 6 | 7 | 13
    White | 13 | 11 | 24
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Syndrome Components
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Melatonin: Cross-over design for subjects on Melatonin for 10 weeks measured at baseline and 10 weeks
- Placebo: Cross-over design for all subjects on Placebo for 10 weeks measured at baseline and at 10 weeks.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 37 | 39
mmHg | -2.7 (11.3) | 4.7 (13.8)
Statistical Analysis 1: Comparison: Melatonin vs Placebo; Average change in systolic blood pressure from pre-treatment baseline to post-treatment at 10 weeks when those subjects were on Melatonin was compared to the average change in systolic blood pressure from pre-treatment baseline to post-treatment at 10 weeks when those same subjects were on Placebo using an intent-to-treat mixed model. Power was estimated based on having 30 subjects completing both the melatonin arm and the placebo arm; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = 6.0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Melatonin First: Cross-over design for subjects randomized to Melatonin First, Placebo Second
- Placebo First: Cross-over design for subjects randomized to Placebo First, Melatonin Second
Arm/Group | Melatonin First | Placebo First
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin First (N=19) | Placebo First (N=20)
Mild stroke (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was designed as a pilot Phase II cross-over design to study the safety of melatonin and to estimate the effect sizes associated with average changes while subjects were on melatonin versus average changes while subjects were on placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes